CLINICAL TRIAL: NCT01897922
Title: The Effects on Growth and Tolerance of an Infant Formula Fed to Term Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mead Johnson Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 3385-2
Record Dates: First submitted 2013-07-03; First posted 2013-07-12 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: Growth of Term Infants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Marketed routine infant formula (Active Comparator)
  Interventions: Other: Control: Marketed routine infant formula
- Infant formula containing a probiotic source (Experimental)
  Interventions: Other: An investigational infant formula containing a probiotic source

INTERVENTIONS:
Other: An investigational infant formula containing a probiotic source
  Arms: Infant formula containing a probiotic source
Other: Control: Marketed routine infant formula
  Arms: Marketed routine infant formula

SUMMARY:
This clinical trial will evaluate an investigational infant formula with a probiotic to determine if it provides normal growth and if it is well tolerated by term infants compared to a marketed routine infant formula.

ELIGIBILITY:
Inclusion Criteria:

* Singleton, 12-16 days of age at randomization
* Term infant with birth weight of a minimum of 2500 grams
* Solely formula fed
* Signed Informed Consent and Protected Health Information

Exclusion Criteria:

* History of underlying metabolic or chronic disease or immunocompromised
* Feeding difficulties or formula intolerance

Ages: 12 Days to 16 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 348 (Actual)
Dates: Start 2013-07; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Body weight measured at each study visit | 3.5 months

SECONDARY OUTCOMES:
Recall of infant formula intake at each study visit | 3.5 months
Body length measured at each study visit | 3.5 months
Recall of stool consistency measured at each study visit | 3.5 months
Medically-confirmed adverse events collected throughout the study period | 3.5 months
Parental Study Product Assessment Questionnaire completed at Study Visit 2 | once
Head circumference measured at each study visit | 3.5 months
Recall of gastrointestinal tolerance measured at each study visit | 3.5 months

CONTACTS AND LOCATIONS:
Overall Officials: Carol Lynn Berseth, M.D., Study Director — Mead Johnson Nutrition
Locations (22):
- United States (22):
  - Birmingham Pediatric Associates, Birmingham, Alabama
  - Greenvale Pediatrics Hoover, Birmingham, Alabama
  - Southeastern Pediatric Associates, Dothan, Alabama
  - Pediatrics East - Alabama Clinical Therapeutics, Pinson, Alabama
  - The Children's Clinic of Jonesboro, P.A., Jonesboro, Arkansas
  - Arkkansas Pediatric Clinic, Little Rock, Arkansas
  - Norwich Pediatric Group, P.C., Norwich, Connecticut
  - Children's Research, LLC, Altamonte Springs, Florida
  - Children's Medical Associations, Plantation, Florida
  - Deaconess Clinical Research, Evansville, Indiana
  - Owensboro Pediatrics, Owensboro, Kentucky
  - Woburn Pediatic Associates, Woburn, Massachusetts
  - Cary Pediatric Center, P.A., Cary, North Carolina
  - Capital Pediatrics & Adolescent Center, Raleigh, North Carolina
  - Pediatric Associates of Mt. Carmel, Inc, Cincinnati, Ohio
  - Pediatric Associates of Fairfield, Inc., Fairfield, Ohio
  - Parma Pediatrics, Inc, Parma, Ohio
  - UHMP Comprehensive Pediatrics, Westlake, Ohio
  - The Jackson Clinic - North Jackson, Jackson, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - Austin Diagnostic Clinic, Austin, Texas
  - DCOL Center for Clinical Research, Longview, Texas

REFERENCES:
- [Derived] Berseth CL, Yeiser M, Harris CL, Kinnaman JN, Lappin V, Wampler JL, Zhuang W, Vanderhoof J. Infant formula with added Lacticaseibacillus rhamnosus GG supported adequate growth and was well tolerated in healthy term infants: a randomized controlled trial. Front Pediatr. 2024 Oct 23;12:1456607. doi: 10.3389/fped.2024.1456607. eCollection 2024. PMID 39507493